CLINICAL TRIAL: NCT06872853
Title: Evaluation of Rare and Complex Tumours of the Thoraco-Abdominal and Soft Tissue District - Observational Study With Retrospective and Prospective Phase
Brief Title: Evaluation of Rare and Complex Tumours of the Thoraco-Abdominal and Soft Tissue District
Acronym: RAC
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RAC - 1058/2020/OSS/AOUBo
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Rare Malignant Neoplasm
MeSH Terms: interventions — Surgical Procedures, Operative; Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: diagnosis, surgery, drugs for rare neoplasms — diagnostic and surgical procedures, drugs (pharmacological active substance, dose, regimen)

SUMMARY:
The goal of this observational study is to collect structured data about diagnosis, treatment and follow-up of rare and highly complex neoplasms.

The study has a rerospective part that will consist in gathering data on patients accessing IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di S. Orsola from 01/01/2000 to 28/09/2017 and a prospective one ranging from 29/09/2017 to 31/12/2025.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologic diagnosis of rare or highly complex malignant neoplasm
* informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients over 18 years of age with a diagnosis of histologically proven rare or highly complex malignant tumour
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2017-09-29 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of different malignant rare neoplasms | Throughout the lenght of study, an average of 10 years
  Description of types of tumours

SECONDARY OUTCOMES:
Response rate (RR) | Throughout the lenght of study, an average of 10 years
  Response rate to different treatments (surgery, drugs)
Local recurrence rate | Throughout the lenght of study, an average of 10 years
  Incidence of local recurrence
Progression-free survival (PFS) | Throughout the lenght of study, an average of 10 years
  Progression-free survival (PFS) assessed for different types of rare malignant neoplasms
Overall survival (OS) | Throughout the lenght of study, an average of 10 years
  OS assessed for different types of rare malignant neoplasms

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Pantaleo, MD, Principal Investigator — Oncology Unit, IRCCS AOUBO
Locations (2):
- Italy (2):
  - Oncology Unit, IRCCS AOUBO Policlinico di S. Orsola, Bologna, BO
  - Thoracic Surgery Unit, Bologna, BO

IPD SHARING:
Plan to Share IPD: No